CLINICAL TRIAL: NCT01843257
Title: Pharmacokinetics and Pharmacological Effects of Alcohol After Bariatric Surgery
Brief Title: Effects of Alcohol After Bariatric Surgery
Acronym: RBA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Missouri-Columbia (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NCT01843257
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: Alcohol intake after bariatric surgery; Alcohol and bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Ethanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Gastric Bypass longitudinal: Morbidly obese subjects undergoing gastric bypass surgery. Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery. The two testing sessions will be repeated ~ 9 months after surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first
- Gastric Banding longitudinal: Morbidly obese subjects undergoing laparoscopic gastric banding surgery. Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery. The two testing sessions will be repeated ~ 9 months after surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first
- Gastric Bypass (cross-sectional): Subjects who underwent gastric bypass surgery 1-5 years ago. Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first
- Gastric Banding (cross-sectional): Subjects who underwent gastric banding surgery 1-5 years ago. Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first
- Sleeve gastrectomy (longitudinal): Morbidly obese subjects who will undergo sleeve gastrectomy. Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery. The two testing sessions will be repeated ~ 9 months after surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first
- Sleeve gastrectomy (cross-sectional): Subjects who underwent sleeve gastrectomy 1-5 years ago. Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first
- No bariatric surgery control: Control group of women with age and BMI similar to those in the cross-sectional arm of the study who have not undergone bariatric surgery.
  Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion before surgery.
  Interventions: Other: Alcohol challenge test Alcohol visit first; Other: Alcohol challenge test Placebo visit first

INTERVENTIONS:
Other: Alcohol challenge test Alcohol visit first — Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion (visit 1 alcohol, visit 2 placebo).
Other: Alcohol challenge test Placebo visit first — Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion (visit 1 placebo, visit 2 alcohol).

SUMMARY:
The investigators wish to study the effects of three forms of bariatric surgery: gastric bypass, sleeve gastrectomy, and lap banding. The surgery is not part of the clinical trial. If insurance does not cover the procedure, then the patient is responsible for payment of the surgical process. The investigators are doing pre- and post-surgery testing to provide a better understanding of the effect of bariatric surgery-induced weight loss on 1) alcohol absorption, distribution and elimination from the body; 2) the effects of alcohol on blood sugar; and 3) the effects of alcohol on mood.

DETAILED DESCRIPTION:
The study includes seven groups of women: One group will be undergoing gastric bypass, another group will be undergoing lap banding, a third group will be undergoing sleeve gastrectomy, the fourth group will be women who underwent gastric bypass 1-5 years ago, the fifth group will be women who underwent lap banding 1-5 years ago, the sixth group will be women who underwent sleeve gastrectomy 1-5 years ago, and the seventh group will be a control group who have not undergone bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Drink alcohol at least once per month

Exclusion Criteria:

* Men
* Drinks more than 7 standard drinks per week or more than 4 standard drinks in a period of 2 hours for the month before enrolling in the study.
* Regular use of drugs of abuse or use of any medication interacting with alcohol pharmacokinetics or pharmacologic effects.
* Alcohol dependence
* Pregnancy, lactation or not using effective methods of birth control
* Smoking
* Anemia
* Liver disease

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bariatric surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change from before bariatric surgery in alcohol's Tmax, Cmax, area under the curve and elimination rates at approximately 9 months after bariatric surgery | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  Time to reach maximum peak blood alcohol levels, alcohol area under the time-concentration curve and alcohol's constant of elimination will be examined before and after surgery and compared between those who had gastric bypass versus lap banding.
Change from before bariatric surgery in alcohol subjective effects at approximately 9 months after bariatric surgery | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  Validated instruments (such as the Addiction Research Center Inventory) will be used to measured alcohol's subjective effects at different timepoints after drinking an alcoholic or a non-alcoholic (control) beverage.

SECONDARY OUTCOMES:
Change from before bariatric surgery on alcohol's effects on glucose homeostasis at approximately 9 months after bariatric surgery | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana Champaign, St Louis, Missouri, United States

REFERENCES:
- [Derived] Pepino MY, Okunade AL, Eagon JC, Bartholow BD, Bucholz K, Klein S. Effect of Roux-en-Y Gastric Bypass Surgery: Converting 2 Alcoholic Drinks to 4. JAMA Surg. 2015 Nov;150(11):1096-8. doi: 10.1001/jamasurg.2015.1884. No abstract available. PMID 26244751